CLINICAL TRIAL: NCT03621254
Title: Investigation Into Optimal FES Training Characteristics After Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-11
Record Dates: First submitted 2018-07-13; First posted 2018-08-08 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Spinal Cord Injury
Keywords: Functional Electrical Stimulation; Exercise Training; Aerobic Fitness; Muscle Strength
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- [HI-SHORT] (Experimental): High-intensity interval training modality of exercise using FES-evoked leg cycling. Three-four times weekly over 6-8 weeks (24 therapy sessions). The programme is 10 x 2-min exercise intervals with 1-2 min of recovery between intervals. High intensity is achieved by high FES current amplitude (120-150 milliampere, patient dependent)
  Interventions: Other: [HI-SHORT
- [LO-LONG] (Active Comparator): Low-moderate intensity continuous training modality of exercise using FES-evoked leg cycling. Three-four times weekly over 6-8 weeks (24 therapy sessions). The programme is 20+ min continuous exercise. Lower intensity is achieved by lower FES current amplitude (< 90-100 milliampere, patient dependent)
  Interventions: Other: [LO-LONG]

INTERVENTIONS:
Other: [LO-LONG] — Both interventions are different modalities of FES-evoked leg exercise, three-four times per week for 6-8 weeks (24 therapy sessions). The comparator intervention ([LO-LONG]) uses 20-40 min (patient state of fitness dependent) of continuous leg exercise of lower intensity.
  Arms: [LO-LONG]
Other: [HI-SHORT — One intervention ([HI-SHORT]) uses a variety of leg exercise interval training of higher intensity for 10 x 2-min intervals.
  Arms: [HI-SHORT]

SUMMARY:
The aim of this study is to investigate two different modalities of functional electrical stimulation (FES) leg exercise in patients with spinal cord injury (SCI). The primary outcomes being compared are 1. FES-induced leg aerobic fitness, and 2. FES-induced leg strength. There will be two FES-leg training groups, and sub-acute patients with SCI will be randomised between the groups - high-short [HI-SHORT] and low-long [LO-LONG]. Both groups (n=10 per group) will exercise on the Hasomed RehaStim™ exercise ergometer for 6-8 weeks, three-four times per week (24 therapy sessions). [HI-SHORT] will perform 10 x 2-min of high-intensity interval training with a recovery of 1-2 min between exercise bouts. [LO-LONG] will perform 20+ min of continuous exercise at a low-moderate exercise intensity. Exercise intensity for [HI-SHORT] and [LO-LONG] will be titrated by neuromuscular stimulation characteristics. The primary outcomes will be assessed before training commences and after 6-8 weeks of training has been completed.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 6-weeks post-trauma after SCI.
* Traumatic and atraumatic spinal cord injuries between C7 and T10
* Participants diagnosed with "motor complete' spinal cord injury American Spinal Injury Association Impairment Scale A and B.
* Age between 18-75 years old.
* Both male and female.
* Have at least 90º bilateral knee flexion.
* Able to perform FES muscle contractions (not FES intolerant).
* Able to follow verbal instructions.

Exclusion Criteria:

* A recent history of trauma to the lower limb.
* Severe or infected pressure sore on weight-bearing skin areas.
* Illness caused by acute urinary tract infection.
* Uncontrolled spasticity or pain.
* History of cardiovascular / cardiorespiratory disease contraindicating exercise.
* Uncontrolled orthostatic hypotension.
* Unhealed decubiti at electrode placement area.
* Recurrent and uncontrolled autonomic dysreflexia.
* Active heterotopic ossification.
* Other peripheral or central neurologic injury.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-01-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Aerobic Fitness | Day 0 to 6 weeks
  Change of Peak Oxygen Uptake - VO2peak (L/min)

SECONDARY OUTCOMES:
Muscle Near Infrared Spectroscopy | Day 0 to 6 Weeks
  Change of resting muscle arterial oxygen saturation (%)
Strength Fitness | Day 0 to 6 weeks
  Change of Peak Power Output (Watts)

OTHER OUTCOMES:
Muscle Volume | Day 0 to 6 weeks
  Changes of muscle volume (L)
Muscle Fatigue | Day 0 to 6 weeks
  Changes of time (sec) until muscle fatigue occurs as defined by fall of Power Output (Watts) to 20% of original value

CONTACTS AND LOCATIONS:
Overall Officials: Glen M Davis, Prof. Dr., Principal Investigator — University of Sydney
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No